CLINICAL TRIAL: NCT00007865
Title: A Phase II Trial of Ifosfamide, Carboplatin, and Etoposide (ICE) Chemotherapy in Combination With Rituximab as Salvage Therapy
Brief Title: Combination Chemotherapy Plus Rituximab in Treating Patients With Recurrent or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 0032-00-FB; P30CA036727 (NIH); NCI-V00-1635 (Registry Identifier: National Cancer Institute)
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Carboplatin; Etoposide; etoposide phosphate; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: rituximab
  Other Names: Rituxan
Drug: carboplatin
  Other Names: Paraplatin
Drug: etoposide
  Other Names: Etopophos, Toposar
Drug: ifosfamide
  Other Names: Ifex

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy combined with rituximab in treating patients who have recurrent or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the chemosensitivity rate in patients with recurrent or refractory non-Hodgkin's lymphoma treated with ifosfamide, carboplatin, and etoposide (ICE) in combination with rituximab.
* Determine whether the addition of rituximab changes the toxicity profile of the ICE chemotherapy regimen in these patients.

OUTLINE: Patients receive rituximab IV on days 1, 8, and 15 and ifosfamide IV over 1 hour, etoposide IV over 2 hours, and carboplatin IV on days 2-4. Treatment continues every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients who are not candidates for autologous stem cell transplantation may receive 1-4 more courses of chemotherapy without rituximab.

Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 19-39 patients will be accrued for this study within 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent or refractory B-cell non-Hodgkin's lymphoma

  o CD20 positive
* Bidimensionally measurable or evaluable disease
* 19 years old and over
* ECOG 0-2 or Karnofsky 70-100%
* Life expectancy at least 3 months
* WBC at least 3,000/mm3
* Granulocyte count at least 1,000/mm3
* Platelet count at least 100,000/mm3
* Bilirubin no greater than 1.5 times upper limit of normal(ULN)
* AST or ALT no greater than 2.5 times ULN
* Creatinine no greater than 1.5 mg/dL
* Fertile patients must use effective contraception
* Concurrent non-steroidal hormonal therapy allowed for non-disease related conditions (e.g., insulin for diabetes)

Exclusion Criteria:

* No myelodysplastic syndrome or chronic myeloid leukemia
* Not pregnant or nursing/negative pregnancy test
* No other prior malignancy except curatively treated basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the cervix
* No active serious infection
* No other concurrent serious medical condition that would preclude study
* No prior bone marrow or peripheral blood stem cell transplantation for non-Hodgkin's lymphoma
* No other concurrent chemotherapy
* No concurrent corticosteroids except transient administration as antiemetic
* No concurrent radiotherapy
* No other concurrent investigational therapy
* No other concurrent antitumor agents

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09-01 (Actual); Primary Completion 2004-03-01 (Actual); Study Completion 2008-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, MD, Study Chair — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Eppley Cancer Center, Omaha, Nebraska, United States